CLINICAL TRIAL: NCT04501094
Title: A Phase II Study of Bintrafusp Alfa (M7824) in Checkpoint Inhibitor Naive and Refractory Subjects With Urothelial Carcinoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Because of the low accrual and the safety concerns we closed the study.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Andrea Apolo, M.D., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 200142; 20-C-0142
Record Dates: First submitted 2020-08-05; First posted 2020-08-06 (Actual); Results first posted 2022-03-22 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-02

CONDITIONS: Urothelial Cancer
Keywords: TGF-Beta; Immune Therapy; PD-L1; Immunocytokine
MeSH Terms: conditions — Camurati-Engelmann Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 1/Arm 1-Treatment with Bintrafusp alfa (M7824) (Experimental): Treatment with Bintrafusp alfa (M7824)
  Interventions: Drug: Bintrafusp alfa (M7824)

INTERVENTIONS:
Drug: Bintrafusp alfa (M7824) — 1200 mg administered intravenous (IV) every two weeks
  Other Names: M7824

SUMMARY:
Background:

Metastatic urothelial carcinoma is lethal and has no cure. Response rates to current treatments are modest. Researchers want to find new strategies to treat the disease. In this study, they will test a drug called Bintrafusp alfa (M7824). The drug is a new immunotherapy that blocks the pathways that cancer cells use to stop the immune system from fighting cancer.

Objective:

To learn if M7824 can help the immune system's ability to fight urothelial cancer.

Eligibility:

People age 18 and older who have urothelial cancer that has spread to other parts of their body and they have been previously treated with chemotherapy or immunotherapy

Design:

Participants will be screened with a medical history and physical exam. They will have blood and urine tests. They will have imaging scans. They will have an electrocardiogram to measure heart function. Their ability to perform their normal activities will be evaluated. They may have a tumor biopsy. They will take a pregnancy test if needed.

Participants will repeat some of the screening tests during the study.

Treatment will be given in a series of 28-day cycles. Participants will get M7824 once every 2 weeks. It is given through an intravenous infusion. For this, a small plastic tube is put into an arm vein. They will get M7824 until their disease gets worse, they have unacceptable side effects, or they decide to stop treatment.

Participants will have a follow-up visit 30 days after treatment ends. Then they will be followed every 12 weeks in the clinic or by telephone/email. Follow-up will last indefinitely.

DETAILED DESCRIPTION:
Background:

* Metastatic urothelial carcinoma is lethal and incurable with a median overall survival of 14 months from diagnosis.
* Immune checkpoint inhibitors targeting the Programmed death-1 (PD-1)/programmed death-ligand 1 (PD-L1) pathway have greatly changed clinical management of metastatic urothelial carcinoma (mUC) improving survival by 3 months in the second-line setting.
* Five PD-1/PD-L1 inhibitors are Food and Drug Administration (FDA)-approved for for second-line metastatic urothelial carcinoma (mUC), two agents for first-line cisplatin-ineligible mUC. However, response rates are modest, ranging from15-20% in the second-line and 24% in the first-line cisplatin-ineligible.
* Therefore, novel strategies are needed to extend benefit of immunotherapy to the remaining approximately 75% of non-responders.
* Higher levels of transforming growth factor-beta (TGF-beta) are associated with immune escape, therapy resistance and poor outcomes in advanced malignancies. Non-responders to anti-PD-1/PD-L1 antibodies have also been found to have increased TGF-beta in the tumor microenvironment.
* Bintrafusp alfa (M7824) is a novel first-in-class bifunctional fusion protein composed of a monoclonal antibody against PD-L1 fused to the extracellular domain of human TGF-beta receptor II (TGFbetaRII), which effectively functions to sequester or "trap" all three TGF-beta isoforms. A phase I study of M7824 (NCT02517398) demonstrated a manageable safety profile and clinical efficacy among patients with heavily pre-treated advanced solid tumors.
* We hypothesize that M7824 is safe and improves outcomes in patients with checkpoint naive or refractory urothelial carcinoma.

Objectives:

-To evaluate the activity of M7824 as determined by objective response rate (ORR) in two metastatic urothelial carcinoma cohorts:

* Cohort 1: Checkpoint inhibitor naive

  * Cohort 1A: cisplatin ineligible
  * Cohort 1B: refractory post-platinum therapy
* Cohort 2: Checkpoint inhibitor previously treated patients

  * Cohort 2A: previously achieved a Complete Response (CR)/Partial Response (PR)
  * Cohort 2B: previously had Stable Disease (SD)/Progressive Disease (PD)

Eligibility:

* Patients must have a histologically confirmed diagnosis of metastatic urothelial cancer.
* Patients may have been previously treated with prior cytotoxic chemotherapy regimen or targeted agent. Patients may have received any number of prior cytotoxic agents.
* 18 years of age or older

Design:

* This is an open label, non-randomized, single arm phase II trial of M7824 in checkpoint inhibitor naive and previously treated patients with urothelial carcinoma of the bladder.
* M7824 (intravenous 1200 mg fixed dose) will be delivered every 2 weeks
* Patients will receive treatment in cycles consisting of 4 weeks.
* A maximum of 75 subjects will be enrolled in this trial.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Ability to understand the purpose of the study, provide signed and dated informed consent, and able to comply with all procedures.
* Male or female patients aged greater than or equal to 18 years of age at time of consent.
* Patients with histologically confirmed diagnosis of urothelial carcinoma of the urinary tract, including the renal pelvis, ureter, bladder, or urethra. Differentiation with variant histologies (e.g. squamous cell differentiated) will be permitted. Mixed histologies are required to have a dominant urothelial/transitional cell pattern.
* Patients must have metastatic disease defined as new or progressive lesions on cross- sectional imaging. Radiological evaluation should occur within 21 days prior to enrollment.
* Patient must have evaluable and measurable disease, per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1.
* Patients may have been previously treated with prior cytotoxic chemotherapy regimen or targeted agent. Patients may have received any number of prior cytotoxic agents.
* Patients may have had prior immunomodulating therapy including therapy targeting the Programmed death-1 (PD-1)/Programmed Cell Death Ligand 1 (PD-L1 axis (cohort 2A and B) but excluding prior treatment with Bintrafusp Alfa (M7824).
* Pre-treatment tissue biopsy and/or archival tissue availability for PD-L1 expression testing is mandatory for enrollment.
* Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to 2
* Required laboratory values reflective of organ function are listed below:

  * Absolute neutrophil count greater than or equal to 1000/microliter
  * Platelets greater than or equal to 75,000 microliter
  * Hemoglobin greater than or equal to 9 g/dL (erythrocyte transfusions are allowed to achieve acceptable Hgb)
  * Aspartate aminotransferase (AST)/Serum glutamic oxaloacetic transaminase (SGOT)/Alanine aminotransferase (ALT)/Serum glutamic-pyruvic transaminase (SGPT) less than or equal to 1.5 institutional upper limit of normal (ULN) with the following exception:

    ---Patients with liver involvement who have AST and ALT less than or equal to 5 ULN may be enrolled.
  * Total bilirubin within normal limits with the following exceptions:

    * Patients with known Gilbert disease who have serum bilirubin level less than or equal to 3 ULN may be enrolled.
    * Patients with tumor liver involvement bilirubin with less than or equal to 3.0 ULN.
  * International normalized ratio (INR) and activated partial thromboplastin time (aPTT) less than or equal to 1.5 ULN

    ---This applies only to patients who are not receiving therapeutic anticoagulation; patients receiving therapeutic anticoagulation (such as low-molecular-weight heparin or warfarin) should be on a stable dose.
  * Creatinine clearance (CrCl) greater than or equal to 30 mL/min/1.73 m^2 (glomerular filtration rate (GFR) may be used in place of CrCl. Creatinine clearance or estimated glomerular filtration rate (eGFR) should be calculated per institutional standard)
* The effects of M7824 on the developing human fetus are unknown. For this reason, women of child-bearing potential and men must agree to use strict and effective contraception (hormonal or barrier method of birth control; abstinence) during treatment and for at least 65 days for women and 125 days for men, after the last dose of M7824 administration. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
* Human immunodeficiency virus (HIV) positive patients are eligible if on stable dose of highly active antiretroviral therapy (HAART), cluster of differentiation 4 (CD4) counts are greater than 350 cells/mm3 and viral load is undetectable.
* Patients with previously treated brain or central nervous system (CNS) metastases are eligible provided that the subjects have recovered from any acute effects of radiotherapy and is not requiring steroids, and any whole brain radiation therapy or any stereotactic radiosurgery was completed at least 2 weeks prior to M7824 administration.
* Hepatitis B virus (HBV) positive patients are eligible-they must have been treated and on a stable dose of antivirals (eg, entecavir, tenofovir, or lamivudine; adefovir or interferon are not allowed) at study entry and with planned monitoring and management according to appropriate labeling guidance.
* Hepatitis C virus (HCV) positive patients are eligible if participants are on active HCV therapy at study entry and on a stable dose without documented clinically significant impaired liver function test or hematologic abnormalities and with planned monitoring and management according to appropriate labeling guidance.
* Cohort 1A Cisplatin Ineligible Specific Inclusion Criteria (first-line for metastatic cisplatin-ineligible):

  * No prior chemotherapy for inoperable locally advanced or metastatic or recurrent Urothelial Carcinoma (UC)

    ---For patients who received prior adjuvant/neoadjuvant chemotherapy or chemoradiation for UC, a treatment-free interval > 12 months between the last treatment administration and the date of recurrence is required in order to be considered treatment naive in the metastatic setting. Prior local intravesical chemotherapy or immunotherapy is allowed if completed at least 4 weeks prior to the initiation of study treatment.
  * Ineligible ("unfit") for chemotherapy or cisplatin-based chemotherapy as defined by any one of the following criteria:

    * Impaired renal function (CrCl > 30 but < 60 mL/min); GFR should be calculated per institutional standard.
    * A hearing loss (measured by audiometry) of 25 decibels (dB) at two contiguous frequencies
    * Grade greater than or equal to 2 peripheral neuropathy (i.e., sensory alteration or paresthesias including tingling)
    * Eastern Cooperative Oncology Group (ECOG) performance score of 2
    * Patient declines chemotherapy after informed discussion with the study doctor
* Cohort 1B Refractory Post-platinum Therapy Specific Inclusion Criteria (second-line for metastatic disease):

  --Disease progression during or following treatment with a platinum-containing regimen for inoperable locally advanced or metastatic urothelial carcinoma or disease recurrence. Examples of regimens include cisplatin + gemcitabine (GC), methotrexate + vinblastine sulfate + doxorubicin + cisplatin (MVAC), and carboplatin + gemcitabine (CarboGem).

  ---Patients who received prior adjuvant/neoadjuvant chemotherapy and progressed within 12 months of treatment with a platinum-containing adjuvant/neoadjuvant regimen will be considered as second-line patients.
* Cohort 2A Checkpoint Inhibitor Previously Treated Patients that Previously Achieved a Complete Response (CR) or Partial Response (PR) Specific Inclusion Criteria:

  --Patients must have been treated with at least one treatment of a PD-1/PD-L1 checkpoint inhibitor for advance or metastatic UC and achieved a complete response or partial response by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria.
* Cohort 2B Checkpoint inhibitor previously treated patients that previously had stable disease (SD) or progressive disease (PD)
* Specific Inclusion Criteria:

  * Patients must have been treated with at least one treatment of a PD-1/PD-L1 checkpoint inhibitor for advance or metastatic UC and had stable disease or a progressive disease by RECIST 1.1 criteria.

EXCLUSION CRITERIA:

* History of allergic reactions attributed to compounds of similar chemical or biologic composition to M7824 investigational agents used in the study.
* Uncontrolled intercurrent illness including, but not limited to, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Symptomatic central nervous system metastasis.
* Subjects unwilling to accept blood products as medically indicated
* Pregnant women are excluded from this study because M7824 is an agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with M7824, breastfeeding should be discontinued if the mother is treated with these agents.
* Patients with any active or recent history of a known or suspected autoimmune disease (with the exception of diabetes type I, vitiligo, psoriasis, or hypo- or hyperthyroid diseases not requiring immunosuppressive treatment) or recent history of a syndrome that required treatment with either systemic corticosteroids (>10 mg daily prednisone equivalent) or immunosuppressive medications. Inhaled steroids and adrenal replacement steroid doses up to 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease.
* Patients with a currently active second malignancy other than non-melanoma skin cancers or cervical carcinoma in situ or incidental organ-confined prostate cancer found on cystoprostatectomy (provided that the following criteria are met: Stage T2N0M0 or lower; Gleason score <= 3+4, prostate-specific antigen (PSA) undetectable). Patients are not considered to have a currently active malignancy if they have completed therapy and are free of disease for >= 2 years and currently do not require systemic therapy.
* Patients who have received or will receive a live vaccine within 30 days prior to the first administration of study intervention. Seasonal flu vaccines that do not contain a live virus are permitted. Locally approved COVID vaccines are permitted.
* Patients having tumor lesion(s) in the liver or chest which are 10 cm or larger.
* Patients previously treated with M7824.
* Patients previously treated with PD-1/PD-L1 checkpoint inhibitors (for Cohorts 1A and 1B only)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2020-10-26 (Actual); Primary Completion 2021-01-19 (Actual); Study Completion 2021-10-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea B Apolo, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data (IPD) recorded in the medical record will be shared with intramural investigators upon request. In addition, all large scale genomic sequencing data will be shared with subscribers to the database of Genotypes and Phenotypes (dbGaP).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely. Genomic data are available once genomic data are uploaded per protocol Genomic Data Sharing (GDS) plan for as long as database is active
Access Criteria: Clinical data will be made available via subscription to Biomedical Translational Research Information System (BTRIS) and with the permission of the study principal investigator (PI).
  Genomic data are made available via the database of Genotypes and Phenotypes (dbGaP) through requests to the data custodians.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2020-C-0142.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1B - Checkpoint Inhibitor Naïve Participants Who Are Refractory Post-platinum Therapy; Cohort 2B - Checkpoint Inhibitor Refractory Participants With Stable Disease or Progressive Disease: Treatment with Bintrafusp alfa (M7824)
  Bintrafusp alfa (M7824): 1200 mg administered intravenous (IV) every two weeks
Period: Overall Study
Arm/Group | Cohort 1B - Checkpoint Inhibitor Naïve Participants Who Are Refractory Post-platinum Therapy | Cohort 2B - Checkpoint Inhibitor Refractory Participants With Stable Disease or Progressive Disease
Started | 1 | 1
Completed | 0 | 1
Not Completed | 1 | 0
Not completed — Death (unrelated to research) | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1B - Checkpoint Inhibitor Naïve Participants Who Are Refractory Post-platinum Therapy | Cohort 2B - Checkpoint Inhibitor Refractory Participants With Stable Disease or Progressive Disease | Total
Number analyzed (Participants) | 1 | 1 | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 0 | 1
  >=65 years | 0 | 1 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.3 (0) | 71.5 (0) | 66.4 (7.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 1 | 1 | 2
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants With an Objective Response Rate (ORR)
Description: The proportion of evaluable patients with objective response rate (ORR) defined as a partial response (PR) or complete response (CR) at the end of treatment with Bintrafusp alfa (M7824). Response was assessed by the Response Evaluation Criteria in Solid Tumors (RECIST)v1.1. Partial response is at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum of diameters. Complete response is disappearance of all target lesions.
Time Frame: From time measurement criteria are met for CR or PR (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented, approximately 3 months.
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Cohort 1B - Checkpoint Inhibitor Naïve Participants Who Are Refractory Post-platinum Therapy | Cohort 2B - Checkpoint Inhibitor Refractory Participants With Stable Disease or Progressive Disease
Number analyzed (Participants) | 1 | 1
Proportion of participants
  Partial Response | 0 | 0
  Complete Response | 0 | 0

2. Secondary Outcome: Number of Participants With Toxicity Grade >1
Description: The number of participants with toxicity grade >1 assessed by the Common Terminology Criteria for Adverse Events (CTCAE)v5.0. Grade 1 is mild, Grade 2 is moderate, Grade 3 is severe, Grade 4 is life-threatening, and Grade 5 is death related to adverse events.
Time Frame: Until confirmed progression, unacceptable toxicity or trial withdrawal, approximately 4 months and 3 days for cohort 1B and 11 months and 17 days for cohort B.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1B - Checkpoint Inhibitor Naïve Participants Who Are Refractory Post-platinum Therapy | Cohort 2B - Checkpoint Inhibitor Refractory Participants With Stable Disease or Progressive Disease
Number analyzed (Participants) | 1 | 1
Participants
  Grade 1 | 1 | 1
  Grade 2 | 1 | 1
  Grade 3 | 1 | 1
  Grade 4 | 1 | 1
  Grade 5 | 0 | 0

3. Secondary Outcome: Number of Participants With Progression Free Survival (PFS)
Description: PFS is defined as the duration of time from start of treatment to time of progression or death, whichever occurs first. Progression was assessed by the Response Evaluation Criteria in Solid Tumors (RECIST)v1.1 and is defined as at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study; and the appearance of one or more new lesions.
Time Frame: From start of treatment to time of progression or death, approximately 6 weeks (first scheduled restaging scan)
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1B - Checkpoint Inhibitor Naïve Participants Who Are Refractory Post-platinum Therapy | Cohort 2B - Checkpoint Inhibitor Refractory Participants With Stable Disease or Progressive Disease
Number analyzed (Participants) | 1 | 1
Participants | 0 | 0

4. Secondary Outcome: Number of Participants That Survived
Description: Here is the number of participants that survived.
Time Frame: Time from treatment to the date of death from any cause, approximately 11 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1B - Checkpoint Inhibitor Naïve Participants Who Are Refractory Post-platinum Therapy | Cohort 2B - Checkpoint Inhibitor Refractory Participants With Stable Disease or Progressive Disease
Number analyzed (Participants) | 1 | 1
Participants | 0 | 1

5. Other Pre Specified Outcome: Number of Participants With Serious and/or Non-serious Adverse Events Assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0).
Description: Here is the number of participants with serious and/or non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Date treatment consent signed to date off study, approximately 4 months and 3 days for cohort 1B and 11 months and 17 days for cohort B.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1B - Checkpoint Inhibitor Naïve Participants Who Are Refractory Post-platinum Therapy | Cohort 2B - Checkpoint Inhibitor Refractory Participants With Stable Disease or Progressive Disease
Number analyzed (Participants) | 1 | 1
Participants | 1 | 1

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately 4 months and 3 days for cohort 1B and 11 months and 17 days for cohort B.
Arm/Group | Cohort 1B - Checkpoint Inhibitor Naïve Participants Who Are Refractory Post-platinum Therapy | Cohort 2B - Checkpoint Inhibitor Refractory Participants With Stable Disease or Progressive Disease
All-Cause Mortality (participants affected / at risk) | 1/1 | 0/1
Serious Adverse Events (participants affected / at risk) | 1/1 | 0/1
Other Adverse Events (participants affected / at risk) | 1/1 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1B - Checkpoint Inhibitor Naïve Participants Who Are Refractory Post-platinum Therapy (N=1) | Cohort 2B - Checkpoint Inhibitor Refractory Participants With Stable Disease or Progressive Disease (N=1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, Death from progressive (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1B - Checkpoint Inhibitor Naïve Participants Who Are Refractory Post-platinum Therapy (N=1) | Cohort 2B - Checkpoint Inhibitor Refractory Participants With Stable Disease or Progressive Disease (N=1)
Anemia (Blood and lymphatic system disorders) | 1 (2) | 0 (0)
Bacteremia (Infections and infestations) | 1 (1) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (2) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (1) | 1 (1)
Oral hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-06-23): https://cdn.clinicaltrials.gov/large-docs/94/NCT04501094/Prot_SAP_000.pdf
  • Informed Consent Form (2021-06-24): https://cdn.clinicaltrials.gov/large-docs/94/NCT04501094/ICF_001.pdf